CLINICAL TRIAL: NCT05998473
Title: Characterization of Dynamic Stability in Normal Pressure Hydrocephalus and Parkinson's Disease
Acronym: HPGAIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Emilie Hutin, Co-director of laboratory, Henri Mondor University Hospital
Other Study IDs: 2023-A01762-43
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hydrocephalus; Parkinson Disease; Walking, Difficulty; Movement Disorders; Gait Ataxia; Diagnoses Disease
MeSH Terms: conditions — Hydrocephalus; Parkinson Disease; Mobility Limitation; Movement Disorders; Gait Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal pressure hydrocephalus: Patients with a diagnosis of normal pressure hydrocephalus and who performed a gait analysis in laboratories
  Interventions: Diagnostic Test: Dynamic stability measurement
- Parkinson's disease: Patients with a diagnosis of Parkinson's disease and who performed a gait analysis in laboratories
  Interventions: Diagnostic Test: Dynamic stability measurement

INTERVENTIONS:
Diagnostic Test: Dynamic stability measurement — The subject is asked to walk 8 meters 3 times: at free speed, at fast speed, and with large steps.

SUMMARY:
This study aims to characterize dynamic stability disorders in two conditions mainly affecting the elderly and with similar walking deficits: hydrocephalus at normal pressure and Parkinson's disease, to provide the most relevant monitoring criteria in usual care.

DETAILED DESCRIPTION:
Walking disorders in normal pressure hydrocephalus are manifested by slowing and ataxic gait, similar to disorders in Parkinson's disease. No studies in the literature have focused on advanced measures of dynamic stability in hydrocephalus at normal pressure, compared to Parkinson's disease, on large samples. The Laboratory of Analysis and Restoration of Movement, located in a Neurorehabilitation Department, provides quantitative data on gait and in particular dynamic stability as part of additional assessments to help patients follow up. Since 2010, people with normal pressure hydrocephalus or Parkinson's disease regularly benefit from these assessments. Retrospective analysis of all these data would help to better characterize motor disorders in hydrocephalus at normal pressure, by discriminating them from those associated with Parkinson's disease. It would lead to the definition of relevant indices to be used for patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient who performed a walking test in the Laboratory Analysis and Restoration of Movement
* Diagnosis of normal pressure hydrocephalus or Parkinson's disease

Exclusion Criteria:

* Levodopa drugs administrated during a delay of 12 hours before walking test
* Presence of an other neurologic disease or of any disease associated with motor disorders in lower limb.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with normal pressure hydrocephalus or Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Coefficient of variation in step length | 30 seconds
  Coefficient of variation in step length during 8-meter comfortable walking test

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Hutin, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Laboratoire Analyse et Restauration du Mouvement, Créteil, France

IPD SHARING:
Plan to Share IPD: No